CLINICAL TRIAL: NCT05543434
Title: Evaluation of The Clinical & Radiographic Parameters in Controlled Type 2 Diabetic Patients Treated With Non-Surgical Periodontal Therapy With & Without Using Hyaluronic Acid Gel
Brief Title: Application of Hyaluronic Acid in Diabetes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Reem Mohammed Ahmed Al-abbadi, dentist, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Reem
Record Dates: First submitted 2022-09-14; First posted 2022-09-16 (Actual); Last update posted 2022-09-21 (Actual); Status verified 2022-09

CONDITIONS: Periodontal Diseases
MeSH Terms: conditions — Periodontal Diseases | interventions — Hyaluronic Acid

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- hyaluronic acid (Experimental): Application of crosslinked HA gel in pockets after subgingival debridement immediately and one week after.
  Interventions: Drug: Hyaluronic acid
- scaling and root planing (Active Comparator): scaling and root planing using ultrasonic scaler and hand instruments.
  Interventions: Drug: Hyaluronic acid

INTERVENTIONS:
Drug: Hyaluronic acid — anti-inflammatory, anti-edematous, osseoinductive.
  Other Names: Gingigel /Germany

SUMMARY:
sub gingival application of hyaluronic acid create great clinical improvement of periodontal pocket treatment.

DETAILED DESCRIPTION:
To clinically and radiographically evaluate the adjunctive effect of the local application of a 0.8% hyaluronan gel in addition to scaling and root planing in treatment of controlled diabetic patients with stage II periodontitis.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* Patient with controlled diabetic type 2 (HgA1C <7) (Mori et al., 2021).
* Periodontitis stage II.
* Periodontitis grade B.
* Pocket depth > 4 mm.
* Smoking ≤ 10 cigarettes/day.
* Cooperative patients able and accept to come for follow up appointments

Exclusion Criteria:

* • The use of antibiotics or anti-inflammatory drugs 1 month prior to the procedure and till the end of 6 months of follow-up.

  * Having surgical therapy or undergoing orthodontic treatment.
  * Ongoing drug therapy that might have an impact on the clinical signs and symptoms of periodontitis.
  * Pregnant and lactation females.
  * Smoking ˃ 10 cigarettes/day.
  * Patients with poor oral hygiene.
  * Any known allergies

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Estimated)
Dates: Start 2022-12-01 (Estimated); Primary Completion 2023-03-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Clinical attachment level gain | 3 months
  Clinical attachment gain by using UNC15 Periodontal probe/ numerical data

SECONDARY OUTCOMES:
Pocket depth reduction | 3 moths
  Pocket depth reduction by using UNC15 Periodontal probe/ numerical data
Bleeding on probing | 3 months
  Bleeding on probing by using UNC15 Periodontal probe/ binary data
Gingival Recession | 3 months
  Gingival Recession by using UNC15 Periodontal probe/ numerical data
Radiographic Evaluation | 3 months
  by using periapical radiograph with standardized acrylic stent

CONTACTS AND LOCATIONS:
Overall Officials: Reem M Alabbadi, BDS, Principal Investigator — master student; Nesma M Shemais, PHD, Study Director — Lecturer of Oral Medicine and Periodontology- faculty of dentistry/Cairo University; Karim F Elsayed, professor, Study Chair — Associate Professor of Oral Medicine and Periodontology, Faculty of Dentistry, Cairo University
Locations (1):
- faculty of dentistry Cairo university, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Al-Abbadi R, Shemais N, Nawwar A, Fawzy El-Sayed KM. Non-surgical periodontal therapy with and without hyaluronic acid gel in type 2 diabetic stage-II periodontitis patients: a randomized clinical trial. BMC Oral Health. 2025 Jul 15;25(1):1166. doi: 10.1186/s12903-025-06485-2. PMID 40665270